CLINICAL TRIAL: NCT07239674
Title: Desiccated Thyroid Extract Combined With Levothyroxine for TSH Suppression Therapy in Intermediate-to-High Risk Differentiated Thyroid Cancer After Surgery: A National Multicenter, Open-Label, Randomized Controlled Trial
Brief Title: Desiccated Thyroid Extract Combined With Levothyroxine for TSH Suppression Therapy in DTC
Acronym: DELTA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: West China Hospital (Other)
Collaborators: West China Tianfu Hospital, Sichuan University (Unknown); Shang Jin Hospital of West China Hospital,Sichuan University (Unknown); Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, China (Unknown); First Affiliated Hospital of Guangxi Medical University (Other); First Affiliated Hospital of Kunming Medical University (Other); Xijing Hospital of Airforce Medical University (Unknown); Sir Run Run Shaw Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Guizhou Medical University (Other); The Second Affiliated Hospital of Kunming Medical University (Other); The Second Affiliated Hospital of Lanzhou University (Unknown); The Fifth People's Hospital of Qinghai Province （Qinghai Province Cancer Hospital) (Unknown); The Affiliated Hospital of Inner Mongolia Medical University (Other); The First Affiliated Hospital of Shanxi Medical University (Other); General Hospital of Ningxia Medical University (Other); Yantai Yuhuangding Hospital (Other); Sun Yat-sen University (Other); Zhongnan Hospital (Other)
Responsible Party: Principal Investigator, Yu Feng, West China Hospital, Sichuan University, West China Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025(1862)
Record Dates: First submitted 2025-11-16; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Intermediate-to-High Risk Differentiated Thyroid Cancer
Keywords: TSH Suppression Therapy; Desiccated Thyroid Extract; Differentiated Thyroid Cancer; Levothyroxine
MeSH Terms: conditions — Thyroid Diseases | interventions — Thyroid (USP); Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal Group (Experimental): Combination therapy with desiccated thyroid extract and levothyroxine (DTE + L-T4) as the TSH-suppressive regimen.
  Interventions: Drug: desiccated thyroid extract (DTE)+levothyroxine (L-T4)
- Control group (No Intervention): Levothyroxine (L-T4) monotherapy as the TSH-suppressive regimen.

INTERVENTIONS:
Drug: desiccated thyroid extract (DTE)+levothyroxine (L-T4) — Desiccated thyroid extract (DTE) is a dry preparation obtained from animal thyroid glands that contains both thyroxine (T4) and triiodothyronine (T3) in an approximately 4:1 ratio, closely matching the physiological hormone profile secreted by the human thyroid. Combining DTE with levothyroxine (L-T4) may overcome current therapeutic bottlenecks. First, L-T4 given in adequate doses provides the major T4-mediated TSH suppression, while the small amount of T3 supplied by DTE acts directly on pituitary thyrotrophs, bypassing impaired DIO2 conversion; this pharmacodynamic synergy yields tighter TSH control, steadier serum levels, and fewer thyrotoxic side-effects. Second, because thyroid-hormone receptor isoforms are differentially expressed across tissues and display distinct T4/T3 affinities, the combination allows finer tuning of thyroid hormone signaling-maintaining adequate tumor suppression while attenuating adverse cardiac and skeletal effects.
  Arms: Experimantal Group

SUMMARY:
The global incidence of Differentiated Thyroid Cancer (DTC) is rising. While surgery followed by TSH suppression is the standard of care, achieving target TSH levels with levothyroxine (L-T4) monotherapy remains challenging, with only 25-70% of intermediate/high-risk patients attaining it within 6-8 months. This therapeutic dilemma stems from three key issues: impaired T4-to-T3 conversion due to DIO2 polymorphisms, the non-physiological hormone ratio of T4 monotherapy, and L-T4's narrow therapeutic window. This often results in an "under- versus over-suppression" paradox, increasing risks of recurrence, atrial fibrillation, and osteoporosis. Combining L-T4 with desiccated thyroid extract (DTE; T4:T3 ≈ 4:1) may overcome these limitations by bypassing DIO2 defects and providing a more physiological hormone profile, thereby potentially improving TSH control while mitigating side effects. Supported by the 2023 Chinese guidelines and our promising pilot data (82% cumulative target attainment at a median of 1.4 months), we propose a two-stage national study: a multicenter cohort study followed by a randomized trial, to generate high-level evidence for this combination therapy in high-risk DTC.

DETAILED DESCRIPTION:
This study is a multicenter, open-label, randomized controlled trial. Stage 1 eligibility: (1) Age ≥ 18 years；(2) Histologically proven DTC after initial surgery (± ¹³¹I)；(3) ATA recurrence risk intermediate (low-intermediate or high-intermediate) or high；(4) On L-T4 monotherapy: TSH above target despite FT4 ≥ 90 % of normal upper limit；(5) Signed informed consent and agreement to follow-up. Stage 2 eligibility: (1) Age 18-70 years (inclusive)；(2) Histologically proven DTC undergoing first-time surgery；(3) ATA recurrence risk intermediate (low-intermediate or high-intermediate) or high；(4) Signed informed consent and agreement to post-operative follow-up. Exclusion criteria: (1) Non-DTC histology; (2) Hyperthyroidism, toxic adenoma, or toxic nodular goiter; (3) Malabsorptive GI disorders (e.g., H.-pylori gastritis, atrophic gastritis, celiac disease) or history of gastric bypass; (4) Hypersensitivity to levothyroxine or desiccated thyroid; (5) Angina, coronary artery disease, tachyarrhythmia, osteoporosis; (6) Concurrent malignancy; (7) Pregnant, lactating, or planning pregnancy within 12 months; (8) Severe COPD, hepatic or renal insufficiency, uncontrolled hypertension or diabetes, or any condition that could bias outcome assessment; (9) Chronic use of psychotropics, systemic glucocorticoids, amiodarone, chemotherapy, iron, thionamides, PPIs, or other drugs interfering with thyroid hormone; (10) Previous exposure to levothyroxine, desiccated thyroid, or T3 preparations; (11) Participation in another clinical trial that could interfere with this study.

Stage 1 prospectively enrolls patients who underwent initial DTC surgery at participating sites, were classified as intermediate or high recurrence risk, subsequently failed to achieve target TSH suppression on L-T4 monotherapy while having FT4 ≥ 90 % of the normal upper limit. The TSH-suppressive regimen is switched to DTE + L-T4, creating a before-and-after self-control study. Stage 2 screens patients scheduled for initial DTC surgery; eligible participants are randomized 1:1 to experimental arm (DTE + L-T4 combination) and control arm (L-T4). The stage 2 target sample size is 446 patients (223 per arm).

Data collection includes: (1) Baseline characteristics: sex, age, BMI, comorbidities (cardiovascular, endocrine, thyroid, etc.), prior neck irradiation; (2) Pre-operative imaging/labs: laryngoscopy, thyroid US, TSH, FT3, FT4, TT3, TT4; (3) Operative data: procedure type, date, extent of lymph-node dissection; (4) Symptom/QoL: ThyPRO-39 questionnaire; (5) hair-pull test for alopecia; (6) Genetics: DIO2 polymorphism; (6) Post-operative plan: initial TSH-suppression dose, first dosing date, RAI administration; (7) Pathology: histology, TNM stage, molecular results, ATA risk stratum. Follow-up at 1, 3, 6, 9, 12 months post-op and 1 month after every dose adjustment: (1) Vital signs, weight, TSH-suppression details; (2) Imaging/labs: thyroid US, TSH, FT3, FT4, TT3, TT4, Tg, TgAb, calcium, 25-OH-VD; (3) Adverse events: cardiovascular, musculoskeletal, neurologic, GI, allergic reactions; (4) ThyPRO-39 and hair-pull test repeated at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Stage 1 eligibility: (1) Age ≥ 18 years；(2) Histologically proven DTC after initial surgery (± ¹³¹I)；(3) ATA recurrence risk intermediate (low-intermediate or high-intermediate) or high；(4) On L-T4 monotherapy: TSH above target despite FT4 ≥ 90 % of normal upper limit；(5) Signed informed consent and agreement to follow-up. Stage 2 eligibility: (1) Age 18-70 years (inclusive)；(2) Histologically proven DTC undergoing first-time surgery；(3) ATA recurrence risk intermediate (low-intermediate or high-intermediate) or high；(4) Signed informed consent and agreement to post-operative follow-up.

Exclusion Criteria:

* (1) Non-DTC histology; (2) Hyperthyroidism, toxic adenoma, or toxic nodular goiter; (3) Malabsorptive GI disorders (e.g., H.-pylori gastritis, atrophic gastritis, celiac disease) or history of gastric bypass; (4) Hypersensitivity to levothyroxine or desiccated thyroid; (5) Angina, coronary artery disease, tachyarrhythmia, osteoporosis; (6) Concurrent malignancy; (7) Pregnant, lactating, or planning pregnancy within 12 months; (8) Severe COPD, hepatic or renal insufficiency, uncontrolled hypertension or diabetes, or any condition that could bias outcome assessment; (9) Chronic use of psychotropics, systemic glucocorticoids, amiodarone, chemotherapy, iron, thionamides, PPIs, or other drugs interfering with thyroid hormone; (10) Previous exposure to levothyroxine, desiccated thyroid, or T3 preparations; (11) Participation in another clinical trial that could interfere with this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 646 (Estimated)
Dates: Start 2025-11-30 (Estimated); Primary Completion 2027-11-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of adequate TSH suppression | 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  Rate of adequate TSH suppression defined as TSH level reaching the preset suppression target. TSH suppression targets follow the 2023 Chinese Guidelines for Thyroid Nodules and Differentiated Thyroid Cancer (2nd edition): during the initial treatment phase (within 1 year after surgery ± ¹³¹I therapy), serum TSH should be < 0.1 mU/L for high-risk patients and 0.1-0.5 mU/L for intermediate-risk patients.
Time to TSH suppression target | 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  Median number of days from treatment initiation to the first measurement meeting TSH suppression criteria.

SECONDARY OUTCOMES:
Thyroid function test | Preoperative, 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  Thyroid function parameters (TSH, FT3, FT4, TT3, TT4) are measured at every follow-up visit to evaluate the physiological stability of hormone replacement.
Symptoms and quality of life related to thyroid dysfunction | Preoperative, 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  THyPRO-39
Assessment of hair-loss severity | Preoperative, 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  Hair-pull test.
Adverse events (AEs) | 1, 3, 6, 9, 12 months postoperative and 1 month after every dose adjustment
  Adverse events (AEs) refer to any unfavorable medical occurrences that develop during the clinical trial, regardless of whether they are related to the investigational medication. They include:
  Thyroid-hormone-excess-related AEs
  * Cardiovascular system: tachycardia, angina, cardiac insufficiency, atrial fibrillation and other arrhythmias.
  * Musculoskeletal system: osteoporosis, fractures, bone pain. Hypersensitivity/allergic reactions
DIO2 polymorphism analysis | Preoperative
  Genomic DNA is extracted from pre-operative blood. The region containing the target SNP is amplified by PCR, digested with a restriction endonuclease, and genotypes are assigned after electrophoresis based on fragment sizes. The data will be used to explore the relationship between DIO2 genotype, TSH-suppression efficacy, and the FT3/FT4 ratio, providing a molecular basis for individualized therapy.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Turner, H.L., van Etten, J., Firth, D. et al. Modelling rankings in R: the PlackettLuce package. Computational Statistics.2020; 35(3): 1027-1057.
- [Result] Fussey JM, Khan H, Ahsan F, Prashant R, Pettit L. Thyroid-stimulating hormone suppression therapy for differentiated thyroid cancer: The role for a combined T3/T4 approach. Head Neck. 2017 Dec;39(12):2567-2572. doi: 10.1002/hed.24926. Epub 2017 Sep 27. PMID 28960722
- [Result] Hao D, Tian L, He H, Zhu C, Guo L, Zhang K, Zhang J. Efficacy and safety of postoperative levothyroxine sodium tablets for improving serum thyroid hormone levels and tumor marker levels in patients with thyroid tumors. Eur J Transl Myol. 2023 Sep 5;33(3):11582. doi: 10.4081/ejtm.2023.11582. PMID 37668013
- [Result] Wang Z, Angell TE, Sun W, Qin Y, He L, Dong W, Zhang D, Zhang T, Shao L, Lv C, Zhang P, Guan H, Zhang H. Analysis of the strategy of LT4 prescribing and TSH monitoring for thyroid carcinoma after lobectomy. Ann Transl Med. 2020 Oct;8(19):1238. doi: 10.21037/atm-20-4890. PMID 33178770
- [Result] Chen W, Li J, Peng S, Hong S, Xu H, Lin B, Liang X, Liu Y, Liang J, Zhang Z, Ye Y, Liu F, Lin C, Xiao H, Lv W. Association of Total Thyroidectomy or Thyroid Lobectomy With the Quality of Life in Patients With Differentiated Thyroid Cancer With Low to Intermediate Risk of Recurrence. JAMA Surg. 2022 Mar 1;157(3):200-209. doi: 10.1001/jamasurg.2021.6442. PMID 34935859
- [Result] Ming J, Zhu JQ, Zhang H, Sun H, Wang J, Cheng RC, Xie L, Li XR, Tian W, Huang T. A multicenter, prospective study to observe the initial management of patients with differentiated thyroid cancer in China (DTCC study). BMC Endocr Disord. 2021 Oct 21;21(1):208. doi: 10.1186/s12902-021-00871-x. PMID 34670546
- [Result] Yavuz DG, Yazan CD, Hekimsoy Z, Aydin K, Gokkaya N, Ersoy C, Akalin A, Topaloglu O, Aydogan BI, Dilekci ENA, Alphan Uc Z, Cansu GB, Ozsari L, Iyidir OT, Olgun ME, Keskin L, Mert M, Can B, Gungor K, Galip T, Canturk Z, Elbuken G, Pekkolay Z, Kutbay NO, Yorulmaz G, Kalkan AT, Unsal YA, Yay A, Karagun B, Bozkur E. Assesment of attainment of recommended TSH levels and levothyroxine compliance in differentiated thyroid cancer patients. Clin Endocrinol (Oxf). 2022 Dec;97(6):833-840. doi: 10.1111/cen.14787. Epub 2022 Jun 12. PMID 35639050
- [Result] Ku EJ, Yoo WS, Lee EK, Ahn HY, Woo SH, Hong JH, Chung HK, Park JW. Effect of TSH Suppression Therapy on Bone Mineral Density in Differentiated Thyroid Cancer: A Systematic Review and Meta-analysis. J Clin Endocrinol Metab. 2021 Nov 19;106(12):3655-3667. doi: 10.1210/clinem/dgab539. PMID 34302730
- [Result] Ringel MD, Sosa JA, Baloch Z, Bischoff L, Bloom G, Brent GA, Brock PL, Chou R, Flavell RR, Goldner W, Grubbs EG, Haymart M, Larson SM, Leung AM, Osborne JR, Ridge JA, Robinson B, Steward DL, Tufano RP, Wirth LJ. 2025 American Thyroid Association Management Guidelines for Adult Patients with Differentiated Thyroid Cancer. Thyroid. 2025 Aug;35(8):841-985. doi: 10.1177/10507256251363120. PMID 40844370
- [Result] Miranda-Filho A, Lortet-Tieulent J, Bray F, Cao B, Franceschi S, Vaccarella S, Dal Maso L. Thyroid cancer incidence trends by histology in 25 countries: a population-based study. Lancet Diabetes Endocrinol. 2021 Apr;9(4):225-234. doi: 10.1016/S2213-8587(21)00027-9. Epub 2021 Mar 1. PMID 33662333